CLINICAL TRIAL: NCT05276466
Title: Assessment of Urinary Polymerase Chain Reaction (PCR) and Next Generation Sequencing (NGS) Technology in the Evaluation and Management of Females With Chronic Bladder Pain and Cystitis-like Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MicroGenDX (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MDX-001
Record Dates: First submitted 2021-11-04; First posted 2022-03-11 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: BPS; IC; NGS; PCR
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): All subject's samples will undergo the same diagnostic test utilizing Polymerase Chain Reaction and Next-Generation DNA Sequencing
  Interventions: Diagnostic Test: Polymerase Chain Reaction and Next-Generation DNA Sequencing

INTERVENTIONS:
Diagnostic Test: Polymerase Chain Reaction and Next-Generation DNA Sequencing — The qPCR Rapid Screening Panel is a quantitative real-time PCR test for bacteria and fungi.
  Next-Generation DNA Sequencing is the Comprehensive Sequencing test will detect virtually all microbial organisms and fungal pathogens that may be present in patient specimens.

SUMMARY:
Real-world clinical practice multicenter study to determine the clinical implications of employing PCR/NGS technology to identify and treat potential urinary pathogens in female participants identified with bladder pain and/or cystitis-like symptoms.

DETAILED DESCRIPTION:
This is a real-world clinical practice multicenter study to determine the clinical implications of employing PCR/NGS technology to identify and treat potential urinary pathogens in female patients identified with BPS and/or CCS symptoms. Eligible subjects will undergo a baseline/screening visit at which time the following will be collected: demographics/history, physical examination, Numerical Rating Scale (NRS) pain (average and maximum), Female Genito-Urinary Pain Index (F-GUPI), Interstitial Cystitis Symptom Index and Interstitial Cystitis Problem Index (ICSI/ICPI), Acute Cystitis Symptom Score (ACSS), and the Short Form -12.v2 Quality of Life Questionnaire (SF-12). MSU and catheterized urine specimens will be collected for urinalysis (UA), standard culture, and PCR/NGS. Subjects will be stratified based on BPS (NIDDK MAPP criteria) or CCS (based on ACSS criteria) symptoms.

Uropathogens detected on PCR/NGS catheterized specimens will be treated with 10 days of PCR/NGS directed antibiotic therapy which will be recommended by a centralized infectious disease consultant. If there are no uropathogenic bacteria in the catheter specimen, the MSU specimen will be used if positive. Prescribing physicians will adjust those recommendations (choice of antibiotic as well as duration of therapy) based on individual patient's history of antibiotic therapy and known allergies and sensitivities. Subjects with negative PCR/NGS findings for potential uropathogens will be treated with 10 days of empiric antibiotic therapy chosen by the investigator from this list b: 1. Trimethoprim sulfamethoxazole, 2. Macrocrystalline nitrofurantoin, 3. Fosfomycin, and 4. Investigator choice. More than one antibiotic may be prescribed if two or more uropathogens are identified. At the discretion of the treating physician with the consent and shared decision making with the patient, a decision may be made to continue antibiotic therapy beyond 10 days if the patient subjectively believes she is responding. In this study, all subjects will be offered antibiotic therapy, either NGS directed or empiric. Fourteen days after beginning antibiotics, the Subjective Global Assessment (SGA), compliance and safety will be determined via phone call. A clinic visit will be scheduled for 14 days after finishing antibiotics for repeat evaluation of symptoms (NRS pain, F-GUPI, ICSI/ICPI, ACSS, SF-12, SGA) and safety. A MSU urine specimen will be collected from all subjects and submitted for PCR/NGS analysis. Subjects who were PCR/NGS negative and failed empiric therapy will be notified that they likely do not have an infection. Primary analyses will be based on the responder rate (SGA responder rate will be the primary efficacy parameter), symptom change based on the other questionnaires, and safety in BPS/CCS subjects treated with PCR/NGS as well as those treated with empiric therapy. A 40% SGA responder rate, where a responder is defined as markedly or moderately improved on the GRA 7-point scale, will be considered a clinically significant impact. A follow-up visit 4 weeks later will collect similar data as collected at the efficacy visit.

ELIGIBILITY:
Inclusion Criteria: Subjects may be included in the study if they have bladder and/or urethral pain and lower urinary tract storage symptoms and only if they meet all of the following criteria at screening/baseline.

1. Subjects are capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in this protocol.
2. Symptomatic subjects with BPS (NIH/NIDDK/MAPP definition) with perceived bladder pain +/- urinary storage symptoms) or symptomatic patients with CCS (chronic UTI definition based on modified ACSS with dysuria)
3. Subjects with previous failure of standard urine culture directed therapy approach, eg. antibiotic treatment based on previous urine culture results (positive, sterile, or nebulous) failed to provide appreciable clinical benefit.
4. Subjects who have experienced a minimum of 3 months of continuous symptoms
5. Subjects who have a minimum average daily bladder pain score of ≥ 3 on a 0-10 NRS scale in the past 3 months
6. Subjects with no antibiotic therapy for the previous 2 weeks
7. Subjects with no UTI supplements including cranberry, d-mannose, high dose vitamin C and Lactobacillus probiotics for the previous 2 weeks.

Exclusion Criteria: Subjects will be excluded from participating in this study if they meet any of the following criteria:

1. Subjects with any of the following confounding conditions: bladder stones, lower ureteric stones, vaginal candidiasis, urethral diverticulum, urinary retention (≥ 300 mL), overactive bladder (ie, urinary urgency secondary to urinary incontinence), or any other condition/disease, which, in the opinion of the investigator, could compromise patient safety or confound the collection or interpretation of study results.
2. Subjects who are pregnant or planning a pregnancy during the study period
3. Subjects with a history of previous urinary diversion procedure with or without bladder removal or bladder augmentation.
4. Subjects with a history of bladder cystoscopy only within 1 month or cystoscopy with bladder biopsy, hydrodistension, fulguration or triamcinolone injection or treatment of Hunner ulcer performed within 3 months prior to Screening.
5. Subjects undergoing active treatment for cancer - urologic (eg bladder) or other - with surgery, radiation or chemotherapy within previous 8 weeks of screening.
6. Subjects with a neurogenic bladder (due to spinal cord injury, stroke, Parkinson's disease, multiple sclerosis, spina bifida, or diabetic cystopathy).
7. Subjects with genital herpes active within 3 months prior to screening.
8. Subjects with a history of gross (visible) hematuria within 1 year prior to screening that has not been evaluated.
9. Subjects who have had major surgery within the past 3 months or has surgery planned during the study period
10. Subjects with a history of alcohol and/or drug abuse that in the investigator's opinion could interfere with the study evaluations or the patient's safety.
11. Subjects catheterized in the past month
12. Subjects that have received antibiotic treatment based on MicroGenDX's NGS results in the prior 12 months
13. Subjects with indwelling ureteral stents
14. Subjects that have received a bladder instillation within the last 4 weeks

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of PCR/NGS directed antimicrobial therapy assessed by the Global Response Assessment (GRA) | 1 year
  GRA is a 7-point descriptive scale in which subjects self-report that degree that their symptoms improved or worsened compared to baseline. The answers available for the subject includes markedly improved, moderately improved, mildly improved, no change, mildly worse, moderately worse, markedly worse. A responder is a subject who reports that compared to baseline their symptoms are moderately or markedly improved. The primary analysis will determine the proportion of subjects who are responders at the efficacy visit.

SECONDARY OUTCOMES:
Safety of PCR/NGS directed antimicrobial therapy by measuring the incidence of Treatment-Emergent Adverse Events by the SAE questionnaire | 1 year
  Determine the safety of employing a PCR/NGS directed antimicrobial therapy strategy in female subjects with BPS and CCS.
concordance | 1 year
  Evaluate concordance of culture results with PCR/NGS findings in this population of women.
Type of sample comparison | 1 year
  Compare the microbiome of midstream and catheterized urine specimens of symptomatic female subjects with BPS and CCS.
Stratification comparison | 1 year
  Compare urinary microbiome of symptomatic population of women stratified based on PCR/NGS positive and PCR/NGS negative subgroups, positive/negative cultures, and BPS and CCS.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Center for Women's Pelvic Health, Los Angeles, California
  - The University of California San Diego Health, San Diego, California
  - Cooper University Health Care, Camden, New Jersey
  - Wake Forest University Baptist Medical Center Urology, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
Currently no plan to share individual data to other researchers.

REFERENCES:
- [Background] Hanno PM, Burks DA, Clemens JQ, Dmochowski RR, Erickson D, Fitzgerald MP, Forrest JB, Gordon B, Gray M, Mayer RD, Newman D, Nyberg L Jr, Payne CK, Wesselmann U, Faraday MM; Interstitial Cystitis Guidelines Panel of the American Urological Association Education and Research, Inc. AUA guideline for the diagnosis and treatment of interstitial cystitis/bladder pain syndrome. J Urol. 2011 Jun;185(6):2162-70. doi: 10.1016/j.juro.2011.03.064. Epub 2011 Apr 16. PMID 21497847
- [Background] Giannantoni A, Bini V, Dmochowski R, Hanno P, Nickel JC, Proietti S, Wyndaele JJ. Contemporary management of the painful bladder: a systematic review. Eur Urol. 2012 Jan;61(1):29-53. doi: 10.1016/j.eururo.2011.07.069. Epub 2011 Sep 9. PMID 21920661
- [Background] Nickel JC, Stephens-Shields AJ, Landis JR, Mullins C, van Bokhoven A, Lucia MS, Henderson JP, Sen B, Krol JE, Ehrlich GD; MAPP Research Network. A Culture-Independent Analysis of the Microbiota of Female Interstitial Cystitis/Bladder Pain Syndrome Participants in the MAPP Research Network. J Clin Med. 2019 Mar 26;8(3):415. doi: 10.3390/jcm8030415. PMID 30917614
- [Background] Nickel JC, Stephens A, Landis JR, Mullins C, van Bokhoven A, Lucia MS, Ehrlich GD; MAPP Research Network. Assessment of the Lower Urinary Tract Microbiota during Symptom Flare in Women with Urologic Chronic Pelvic Pain Syndrome: A MAPP Network Study. J Urol. 2016 Feb;195(2):356-62. doi: 10.1016/j.juro.2015.09.075. Epub 2015 Sep 26. PMID 26410734
- [Background] Alidjanov JF, Naber KG, Pilatz A, Wagenlehner FM. Validation of the American English Acute Cystitis Symptom Score. Antibiotics (Basel). 2020 Dec 19;9(12):929. doi: 10.3390/antibiotics9120929. PMID 33352734
- [Background] O'Leary MP, Sant GR, Fowler FJ Jr, Whitmore KE, Spolarich-Kroll J. The interstitial cystitis symptom index and problem index. Urology. 1997 May;49(5A Suppl):58-63. doi: 10.1016/s0090-4295(99)80333-1. PMID 9146003